CLINICAL TRIAL: NCT04613180
Title: Effectiveness of Montelukast in Children With Recurrent Obstructive Bronchitis
Brief Title: Evaluation of the Effectiveness of Montelukast in Children With Recurrent Obstructive Bronchitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGU 20170692
Record Dates: First submitted 2020-10-07; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Bronchiolitis
Keywords: Montelukast sodium; Prevention; Relapse; Obstructive bronchitis
MeSH Terms: conditions — Recurrence | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into 2 groups. I the group (control) included 40 patients who received standard therapy. The second group included 40 patients who received oral montelukast sodium. The therapeutic dosage of the drug was 0.2 mg/kg/day, the daily dose was prescribed once a day for the entire duration of the disease. As a prevention of repeated episodes of bronchial obstructive syndrome, the drug was prescribed at a dose of 0.1 mg/kg/day, the duration of anti-relapse therapy was 30 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (control group) (Placebo Comparator): 40 patients with obstructive bronchitis who received placebo
  Interventions: Drug: Placebo
- Group II (Active Comparator): 40 patients who received oral montelukast sodium oral, at a dosage of 0.2-0.4 mg/kg/day
  Interventions: Drug: Montelukast Sodium

INTERVENTIONS:
Drug: Montelukast Sodium — Montelukast is used to prevent wheezing, difficulty breathing, chest tightness, and coughing caused by asthma in adults and children 12 months of age and older. Montelukast is also used to prevent bronchospasm (breathing difficulties) during exercise in adults and children 6 years of age and older.
  Other Names: Singulair
  Arms: Group II
Drug: Placebo — placebo containing no active substance
  Arms: Group I (control group)

SUMMARY:
The aim of the study was to evaluate the effectiveness of montelukast sodium in the treatment and prevention of recurrent obstructive bronchitis in children. The investigators examined 80 children aged 1 to 7 years with recurrent obstructive bronchitis, who were randomly divided into 2 groups.

DETAILED DESCRIPTION:
The aim of the study was to evaluate the effectiveness of montelukast sodium in the treatment and prevention of recurrent obstructive bronchitis in children. The investigators examined 80 children aged 1 to 7 years with recurrent obstructive bronchitis, who were randomly divided into 2 groups. Group I (control) included 40 patients who received standard therapy and placebo. Group II (main) included 40 patients who received standart therapy and oral montelukast sodium.

ELIGIBILITY:
Inclusion Criteria:

* RDA score=6 points
* E:I index score >1.40
* ineffective treatment at home for ≥48 hours
* adverse comorbidities

Exclusion Criteria:

* chronic or congenital diseases of the Central nervous, cardiovascular and bronchopulmonary systems

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of oral administration of montelukast sodium in comparison with placebo in children with obstructive bronchitis | up to 24 months
  Children aged 1 to 7 years with recurrent obstructive bronchitis who will be treated in the Emergency Pediatrics and pediatric intensive care departments of the Emergency hospital of Samarkand will be examined. Patients will be randomly divided into 2 groups. Group I (control) will include 40 patients who received standard therapy and placebo. Group II will include 40 patients who received oral montelukast sodium in addition to standard therapy. Modified bronchophonography will be used to determine the effectiveness of the therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samarkand State Medical Institute, Samarkand, Uzbekistan

IPD SHARING:
Plan to Share IPD: No